CLINICAL TRIAL: NCT01846819
Title: Factors Associated With End Stage Liver Disease
Status: Terminated | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 11-00843
Record Dates: First submitted 2013-05-01; First posted 2013-05-03 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Cirrhosis; Hepatic Encephalopathy; Fatigue; Depression
MeSH Terms: conditions — Fibrosis; Hepatic Encephalopathy; Fatigue; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Ambulatory cirrhotic patients: Severity of liver disease will be assessed through a detailed clinical examination of ascites grade, history of complications from cirrhosis (hepatic coma, spontaneous bacterial peritonitis, gastrointestinal bleeding), laboratory tests (TBili, Albumin, INR, hemoglobin).
  Depression will be assessed with the following questionnaires: Beck Depression Inventory (BDI), EQ-5D, Psychological General Well-Being Index (PGWBI), LDQOL.
  Fatigue will be assessed with the FIS and 6 Minute Walk Test.
  Hepatic Encephalopathy will be assessed with the number connection, digit-symbol coding and inhibitory control test.

SUMMARY:
100 ambulatory cirrhotic patients attending a liver transplant clinic will undergo a comprehensive clinical evaluation for severity of liver disease, anemia, depression, and fatigue. Fatigue will be assessed with the FIS and sub-maximal exercise capacity with the 6-minute walk test (6MWT), a standardized exercise test that measures the distance that a patient is capable of walking in 6 minutes (6MWD). Depression will be assessed by using three well-known questionnaires. The SF-36, Beck's Depression Inventory (BDI-II), EQ-5D, and the Psychological General Well-Being Index (PGWBI). Univariate analysis will be performed to select the factors that potentially are associated with the scores as indicated by a P value <.20; the selected factors will then be entered in a stepwise regression to create a multivariate model giving the combination of factors that are significantly associated with the measure of fatigue and depression. Hemoglobin (Hb) levels will then be added to the model in order to test its significance while controlling for the other factors.

DETAILED DESCRIPTION:
100 ambulatory patients with cirrhosis will be prospectively evaluated for severity of liver disease, anemia, and fatigue; exclusion criteria includes chronic renal insufficiency and recent alcohol use, gastrointestinal bleeding, and infection.

Patients will first be identified and be asked to partake in the study. They will be asked to read over an informed consent form. Subsequently, they will be asked to fill out a depression questionnaire before performing the 6MWT. During the 6MWT the patient will be walking up and down two designated points 100 feet apart. They will be asked to walk for 6 minutes using any walking aids and resting as needed. Their final distance will be recorded. They will then be asked to fill out the FIS fatigue questionnaire.

Severity of liver disease will be assessed through a detailed clinical examination of ascites grade, hepatic encephalopathy, history of complications from cirrhosis (hepatic coma, spontaneous bacterial peritonitis, gastrointestinal bleeding), standard liver tests (TBili, Albumin, INA), platelet count as a parameter of splenic sequestration and portal hypertension, Child-Pugh score, MELD (Model of End-stage Liver Disease) score. Anemia will be assessed with hemoglobin levels. Depression will be assessed with the following questionnaires: Beck Depression Inventory (BDI), EQ-5D, Psychological General Well-Being Index (PGWBI), LDQOL. Fatigue will be assessed with the FIS and 6 Minute Walk Test. Hepatic Encephalopathy will be assessed with the number connection, digit-symbol coding and inhibitory control test. Sexual function will be assessed by the Sexual Problems and Sexual Function scales of the LDQOL. The results will be scored and compared to depression quality of life, and end-stage liver disease factors.

ELIGIBILITY:
Inclusion Criteria:

* male or female, age b/w 18-70 years, inclusive
* willingly and able to provide written consent
* Diagnosed with Cirrhosis
* Able to read and write in English

Exclusion Criteria:

* Inability to provide consent
* Not within age range of 18-70 years, inclusive
* Not diagnosed with Cirrhosis
* Unable to read or write in English
* Unable to walk

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients experiencing cirrhosis of the liver
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2012-07; Primary Completion 2014-05 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Fatigue | 20 minutes
  Patients undergo 6 minute walk test and complete Fisk Impact Scale (Fatigue Questionaire)

SECONDARY OUTCOMES:
Hepatic Encephalopathy | 20 minutes
  Patients do psychometric tests (Number Connection Test, Symbol Digit Coding Test, and Inhibitory Control Test)
Depression | 5 min
  Patients complete Beck Depression Inventory Questionnaire
Quality of Life | 10 min
  Patients complete several questionaires (Liver disease quality of Life, EQ-5D, Psychological Well-Being index)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Sigal, M.D., Principal Investigator — NYU Langone Medical Center
Locations (1):
- NYU School of Medicine, Schwartz Health Care Center Suite 4C, New York, New York, United States